CLINICAL TRIAL: NCT03005431
Title: Parents of Newly Diagnosed Preschool Children With Autism Spectrum Disorder: The Effectiveness of a Self-Directed On-line Parent Training and Support Program on Parent and Child Outcomes
Brief Title: Parents of Newly Diagnosed Preschool Children With Autism Spectrum Disorder:
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, ARobson, Principal Investigator, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HS20295 (H2016:427)
Record Dates: First submitted 2016-12-20; First posted 2016-12-29 (Estimated); Last update posted 2017-10-03 (Actual); Status verified 2017-09

CONDITIONS: Autism
Keywords: Parenting; Training; Support; On-line; Stress
MeSH Terms: conditions — Autistic Disorder | interventions — Palliative Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Parent training and support (Experimental): Parents will be given access to participate in an on-line support forum and a set of on-line parent training modules.
  Interventions: Behavioral: Parent training and support
- Waitlist control group (No Intervention): These parents will receive regular or typical services

INTERVENTIONS:
Behavioral: Parent training and support — Parents will be given access to participate in an on-line support forum and a set of on-line parent training modules.
  Arms: Parent training and support

SUMMARY:
Manitoba parents of preschool children newly diagnosed with Autism must wait up to a year to receive government funded services for their child. During this delay parents need support and training to promote their child's development. The purpose of this research is to develop and evaluate an on-line, parent training and support program that will assist parents during this time. It is predicted that if parents receive on-line training and support they will increase their parenting knowledge and skills, reduce their stress, and create better outcomes for their child, in comparison to parents who do not receive the training. The experimental study (n=60) will use a randomized, masked, waitlist control design that compares a treatment group to a control group. Descriptive statistics will be used to describe differences between groups, ANCOVA's to test for differences between groups, and Pearson correlations to describe the relationship between parent stress and outcomes.

DETAILED DESCRIPTION:
Statement of the Research Problem/Purpose/Objectives Autism Spectrum Disorder (ASD) is a neurological disorder that causes complex developmental difficulties within the first three years of life. Preschool children diagnosed with ASD typically have pervasive deficits in social interaction and communication, and the occurrence of repetitive and restrictive behaviours. Parenting a preschool child with these characteristics, coupled with the devastating impact of their child receiving a diagnosis of ASD, creates high levels of parental anxiety, stress, depression, and general mental health difficulties. Given the seriousness of the child's diagnosis and the compromise in parenting and family functioning, families are referred to formalized treatment programs that provide support for both the child and parents. However, with the recent rise in Autism prevalence rates Manitoba parents now wait up to a year to receive formalized government funded treatment services for their child and family. This delay in formalized service has critically important consequences for the child, the family, and society.

To bridge this gap in service, parents could be afforded the opportunity to participate in a cost efficient self-directed online training and support program specific to parents in Manitoba. Given that there is consistent evidence to support the effectiveness of parent training and involvement once a child has entered a formalized treatment program, the potential effectiveness of parent training and support while waiting for a formalized treatment program should also be considered.

Research on the efficacy and effectiveness of on-line self-directed Autism parent training programs is extremely limited. Additionally, there is a lack of knowledge regarding the appropriate content, timing, and duration of a training program for parents of newly diagnosed children with ASD and conflicting evidence on the interactional effects between parent training and levels of parenting stress during this time period.

The primary purpose of this study is to address the training and support requirements of parents of preschool children newly diagnosed with ASD, by developing and evaluating the effectiveness of a self-directed on-line ASD parent training and support program. The secondary purpose is to assess the interactional effects, of a self-directed on-line ASD parent training and support program, and parent stress, on parent and child outcomes. It is predicted that if parents receive on-line training and support they will increase their parenting knowledge and skills, reduce their levels of stress, and create better engagement and communication outcomes for their child, in comparison to parents who do not receive the training and support.

Methods: The experimental study will use a randomized, masked, waitlist control design that compares an intervention treatment group to a waitlist control group. After meeting criteria and consent requirements for participation in the study, all families will participate in pre-measures. Families will then be randomized to either a treatment group or a waitlist control group. After pre measures the treatment group parents will receive access to the on-line self-directed training and support program for a 4-month period. After this time period both groups will then be re-assessed on the Parent and Child outcome measures and then the Waitlist Group will be given access to the on-line self-directed training and support program.

Procedure. After a family has been assessed as eligible for the study, and have signed consent forms to participate in the study, they will be given an appointment time to attend the nursery setting for pre-measures. One parent will be asked to engage in free play with their child similar to how they would at home (using a standardized set of toys). The parent will be video recorded playing with their child for a ten-minute period, and then asked to answer the three questionnaires. This procedure will occur at baseline (Time 1, within 2 months of diagnosis), and after the treatment period (Time 2, at least four months after the baseline measure). After base-line measures, families will be randomly assigned to the treatment group, and the waitlist group, using a random numbers table and a pre-arranged opaque envelope system. Treatment group parents will then be given access to participate in the on-line self-directed parent training and support intervention between Time 1 and Time 2, and the waitlist group parents will be given access to the intervention after Time 2. Parents will be given codes to access the on-line resources to ensure their anonymity to other participants. The codes will also allow the principle investigator to track when parents access the on-line training and support and when they have completed the on-line training. When treatment group parents have completed the on-line training (and after at least a four-month period has elapsed since the baseline measure) the parent and child will be invited back to the nursery setting for Time 2 measurements.

Additionally, after a four-month period the matched waitlist group parent and child will be invited back to the original setting for Time 2 measurements, after which they will be given access to the on-line training and support. Families that signed consent forms and then dropped out, will also be given access to the on-line training and support, at this time. The personnel used to administer, score and input the data for the questionnaires, and observational measures, will be masked as to the participant's group assignment and time of measure. All data will contain only the code with no specific participant identifiers. All digital video recordings, questionnaires, observations sheets, and participant code sheets will be kept in a locked cabinet in the office of the main investigator and on a password protected secured government server. Inter-observer agreement will be used in the observation measures of the parent's intervention techniques and the child's measures of engagement and communication. For these observational measures, personnel will be trained by the primary investigator. Inter-observer agreement will be used in a training procedure until personnel meet or exceed 80% agreement on each measure for two consecutive observation trials. Additionally, after all observation data has been collected, a random sample of 20% of the data for each measure will be scored by two personnel, and inter-observer agreement will be reported.

The independent variable is the on-line self-directed parent training and support program. Each on-line module contains multi-media presentations (written material, graphics, and video's), links to additional materials found on the internet, summaries of key information, small quizzes that help parents focus on important material and an accompanying parent workbook. In addition, parents are directed in Module 2 to an on-line parenting support and information sharing forum exclusive to the parents in the training program. Through the on-line forum parents can access a professional autism specialist and other parents involved in the study, and are able to ask questions, answer questions, provide comments, discuss issues, and in general receive support and give support to others.

Four specific hypotheses will be tested for statistical significance. The first hypothesis is: Parents in the treatment group will have significantly higher Family Support, Knowledge and Intervention Techniques scores, and significantly lower Stress scores at Time 2, compared to the control group. This hypothesis will be tested individually for each measure using an Analysis of Covariance design (ANCOVA) to test for differences between groups while adjusting for any initial difference.

The second hypothesis is: Children of parents in the treatment group will have significantly higher scores in Engagement and Communication at Time 2 compared to children of parents in the control group. This hypothesis will be tested individually for each measure using an Analysis of Covariance design (ANCOVA) to test for differences between groups while adjusting for any initial difference.

The third hypothesis is: Parent's perceived level of stress will moderate the treatment effects on Parent outcomes measures of Knowledge and Intervention Techniques at Time 2. Specifically, it is hypothesized that there will be a negative (inverse) correlation between Parent stress scores at Time 1 and Parent Knowledge and Intervention Technique scores at time 2 (the higher the parent's stress score at Time 1, the lower the parent's Knowledge and Intervention Technique scores at Time 2). Additionally, it is hypothesized that there will be a negative (inverse) correlation between the parent's change in stress scores from Time 1 to Time 2 to parent's Knowledge and Intervention Technique scores at Time 2 (as parents perceived level of stress decreases from Time 1 to Time 2 parent's Knowledge and Intervention Technique scores will increase at Time 2). Correlations will be conducted using Pearson's product-moment (r) calculations.

The fourth hypothesis is: Parent's perceived level of stress will moderate the treatment effects on Child outcomes measures of Engagement and Communication at Time 2. Specifically, it is hypothesized that there will be a negative (inverse) correlation between Parent stress scores at Time 1 and Child Engagement and Communication scores at time 2 (the higher the parent's stress score at Time 1, the lower the Child Engagement and Communication scores at Time 2). Additionally, it is hypothesized that there will be a negative (inverse) correlation between the parent's change in stress scores from Time 1 to Time 2 to the Child's Engagement and Communication scores at Time 2 (as parents perceived level of stress decreases from Time 1 to Time 2 the Child's Engagement and Communication scores will increase at Time 2). Correlations will be conducted using Pearson's product-moment (r) calculations.

Process for Seeking Consent Initial screening for patients that meet the criteria will be done by the Developmental Pediatricians at the Child Development Clinic. When patients are in the SSCY Centre for a counsel with their Pediatrician, the Pediatrician will provide the families of all those who meet the inclusion criteria with a study advertisement containing the PIs contact information. Parents who phone the Principal Investigator to find out more about their participation in the study will be given the option of meeting the Principal Investigator at an office in the SSCY Centre or at their home, or at a place of their choosing. The Principal Investigator will explain the study and the consent form at that time. Parents will be told that they do not need to decide immediately and that they have the option of reviewing the study documentation and consent forms with others, and at their convenience. They will also be given a phone number to call if they have any further questions.

ELIGIBILITY:
Inclusion Criteria:

Children will be eligible for the study if they are less than 60 months of age and have a formal documented diagnosis of ASD.

Exclusion Criteria:

* Children who have another formally diagnosed co-morbidity (e.g. Cerebral Palsy, FASD, ADHD), or who have parents not able to read English will be excluded from the study.

Max Age: 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Change in the Parent's Knowledge of ASD and Early Home Intervention Questionnaire. | Baseline and then in four months
  This questionnaire was developed specifically for this study to assess the parent's perceptions of their knowledge of ASD and early home intervention techniques. This questionnaire was developed because no pre-existing measure could be found that addressed caregiver perceptions of their knowledge of ASD and early intervention techniques. Parents in the study will respond to 30 questions related to the diagnosis of ASD (e.g. I understand how ASD is diagnosed.); characteristics of children with ASD (e.g. I understand why my child may have unusual sensory interests); parental support (e.g. I know the services available in the community to support my child and family); and parent early intervention techniques (e.g. I know ways to promote communication in my child) using a 5 point scale from 1 (no understanding) to 5 (an excellent understanding) to produce an overall score (range 30 to 150).
Change in the Early Intervention Techniques Parent Rating Scale. | Baseline and then in four months
  This rating scale assesses the parent's use of early intervention techniques during the pre and post 10 minute video recorded parent/child play session. The rating scale was developed specifically for this study to assess the parent's use of the early intervention techniques specific to the training involved in this study. The examiner will watch the ten minute video and then rate the parents on their frequency of usage of seven early intervention techniques; 1) Follows the Child's Lead/Engages Child, 2) Imitation, 3) Expanding/Modelling, 4) Reciprocity/Turn Taking, 5) Promotes Communication, 6) Promotes Regulation, and 7) Promotes Appropriate Behaviour. Each individual item is rated using 1-5 Likert scale for frequency, 1) Never, 2) Rarely, 3) Sometimes, 4) Often, 5) Always, to produce an overall score (Range 7-35).
Change in Parent/Child Joint Engagement | Baseline and then in four months
  An observational measure will be used to evaluate the child's level of joint engagement with the parent during the pre and post 10 minute video recorded parent/child play session. An evaluation of joint engagement was chosen as it is an important metric of parent child interactions, an important developmental precursor to communication, and a measurement that has been shown to be sensitive to treatment related changes for toddlers and early preschool children (Kasari et al., 2010; Schertz, Odem, Baggett, & Sideris, 2013). The 10 minute parent/child video recorded play session from both pre and post intervention will be observed continuously and coded in 5 second intervals for three levels of child engagement: Unengaged, Object Engagement, and Joint Engagement. A data collection sheet for the time sampling procedure will be used to record a 120 - 5 second intervals, which will total 10 minutes.
Change in Expressive Communication Measure | Baseline and then in four months
  An observational measure will be used to evaluate the child's expressive communication during the pre and post 10 minute video recorded parent/child play session. An expressive communication measure was chosen because it is a core deficit of ASD and a common outcome measure used to evaluate parent training interventions for toddlers and preschoolers with ASD (Beaudoin, Sebire, & Couture, 2014). The 10 minute parent/child video recorded play session from both pre and post intervention will be observed continuously and coded in 5 second intervals for five levels of child expressive communications: Gestures, Vocalizations, Word approximations, Words, and Multi-word utterances. Operational definitions from Harjuson-Webb and Robbins, (2012), are used. A data collection sheet will be used to record a frequency count in each category over the 10 minute video recorded caregiver/child play session.

SECONDARY OUTCOMES:
Change in the Parenting Stress Index-Short Form | Baseline and then in four months
  The PSI-SF was chosen because it is a widely-used instrument for measuring parent stress with a variety of parent groups including parents of children with autism (Zaidman-Zait, et al., 2011). Parent's respond to 36 items (e.g. "I feel trapped by my responsibilities as a parent." "I feel alone and without friends.") using a five point scale from 1 (strongly agree) to 5 (strongly disagree). All 36 items are then reverse scored with a final higher score indicating a higher level of stress. The overall score (range 36-180) of parent stress is produced, as well as three subscale scores; Parental Distress (PD), Parent-Child Dysfunctional Interaction (P-CDI), and Difficult Child (DC). The short form is correlated to the full length PSI at .94 and has an internal consistency coefficient alpha of .91 for the total scale, .87 for (PD), .80 for (P-CDI), and .85 for (DC); and a test-retest reliability coefficient of .84 for the total scale, .85 for (PD), .68 for (P-CDI), and .78 for (DC).
Change in the Family Support Scale | Baseline and then in four months
  The FSS was chosen to identify and quantify the sources of the parent's social support network pre and post intervention. Parents respond to 18 items (e.g. My Friends, Co-workers, Day Care, Other parents, etc.) in regards to a single question, "How helpful has each of the following been to you in terms of raising your child?" Parent's respond by using a five point scale from 0 (Not available) to 5 (Extremely helpful) to produce a total overall score (Range 0 - 90). The Scale has an internal coefficient alpha of .79, and a test-retest reliability coefficient of .91 (Dunst, Jenkins, & Trivette, 1984).

CONTACTS AND LOCATIONS:
Overall Officials: Andrew T Robson, M.Sc., Principal Investigator — University of Manitoba

IPD SHARING:
Plan to Share IPD: No